CLINICAL TRIAL: NCT00720564
Title: A Phase I Study of the Combination of Radiation Therapy (RT), Arsenic Trioxide (ATO) and Temozolomide (TMZ) in Patients With Newly-Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: Radiation Therapy, Arsenic Trioxide, and Temozolomide in Treating Patients With Newly Diagnosed High-Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Jana Portnow, City of Hope Comprehensive Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000600335; P30CA033572 (NIH); CHNMC-07058; CEPHALON-CHNMC-07058
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult gliosarcoma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma; Glioma | interventions — Arsenic Trioxide; Temozolomide; Chemotherapy, Adjuvant; Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide
Drug: temozolomide
Procedure: adjuvant therapy
Radiation: intensity-modulated radiation therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as arsenic trioxide and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Arsenic trioxide and temozolomide may also make tumor cells more sensitive to radiation therapy. Giving radiation therapy together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of arsenic trioxide when given together with temozolomide and radiation therapy in treating patients with newly diagnosed high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of arsenic trioxide when administered sequentially with temozolomide during radiotherapy in patients with newly diagnosed glioblastoma multiforme.
* Determine the dose-limiting toxicities of this regimen in these patients.

OUTLINE: This is a dose-escalation study of arsenic trioxide.

Patients undergo radiotherapy (may be intensity-modulated) on days 1-5. Patients also receive arsenic trioxide IV over 1-2 hours on days 1-5, and oral temozolomide on days 1-7. Treatment with radiotherapy, arsenic trioxide, and temozolomide repeats every week for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients may then receive oral temozolomide on days 1-5. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed grade III or IV glioma including any of the following:

  * Glioblastoma
  * Anaplastic astrocytoma
  * Gliosarcoma
  * Anaplastic oligodendroglioma
  * Anaplastic oligoastrocytoma
* Measurable or nonmeasurable disease
* No more than 5 weeks since prior brain surgery

  * Recovered from surgery, post- operative infection, and other complications
* Preoperatively and postoperatively diagnostic contrast-enhanced MRI or CT scan of the brain performed prior to radiation therapy

  * Patients diagnosed by stereotactic biopsy do not require the postoperative scan

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 60%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 mg/dL
* AST ≤ 4.0 times ULN
* No prolonged QT interval > 460 milliseconds on baseline electrocardiogram in the presence of normal serum potassium and magnesium
* No uncontrolled electrolyte imbalance (i.e., sodium < 132 mmol/L, potassium < 3.5 mEq/dL, magnesium < 1.7 mg/dL)
* No history of torsades de pointes type of ventricular arrhythmia
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No medical or psychiatric illness that, in the investigator's opinion, could potentially preclude the completion of study therapy
* No HIV positivity
* No active connective tissue disorders (e.g., lupus or scleroderma) that, in the investigator's opinion, may put the patient at high risk for radiation toxicity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior brain radiotherapy or chemotherapy for brain tumor
* Concurrent corticosteroids to control cerebral edema allowed provided dose is stable or decreasing for the past 5 days
* No concurrent or plan to receive drugs that are known to prolong the QT interval
* No prior radiation to the head or neck (except for T1 glottic cancer) resulting in overlap of radiation fields

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of arsenic trioxide
Dose-limiting toxicities as measured by CTCAE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States